CLINICAL TRIAL: NCT01015651
Title: Assessment of the Nociception During Lumbar Surgery
Acronym: CARDEAN-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Jean-Francois PAYEN, Anesthesia and Intensive Care, University Hospital, Grenoble
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 0823; 2008-A01602-53 (Registry Identifier: ID RCB)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2010-04-07 (Estimated); Status verified 2010-04

CONDITIONS: Lumbar Surgery
Keywords: nociception, intraoperative, baroreflex
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- remifentanil-2 (Active Comparator): In this group, patients are receiving a continuous i.v. infusion of remifentanil according to a target effect site concentration of 2 ng/ml.
  Interventions: Drug: remifentanil
- remifentanil-4 (Active Comparator): In this group, patients are receiving a continuous i.v. infusion of remifentanil according to a target effect site concentration of 4 ng/ml.
  Interventions: Drug: remifentanil

INTERVENTIONS:
Drug: remifentanil — anesthesia is induced and maintained with a target-controlled infusion of remifentanil at 2 ng/ml.
  Arms: remifentanil-2
Drug: remifentanil — anesthesia is induced and maintained with a target-controlled infusion of remifentanil at 4 ng/ml.
  Arms: remifentanil-4

SUMMARY:
The aim of the study is to assess the accuracy of a new paradigm in measuring the level of nociception during lumbar surgery. The paradigm is based the measurement of the baroreflex in response to noxious stimuli in anesthetized patients.

DETAILED DESCRIPTION:
The study aims at exploring the changes in the baroreflex induced by 3 noxious stimulation in anesthetized patients: tracheal intubation, tetanic stimulus, and surgical incision. Patients are randomly assigned to one of 2 groups: remifentanil-2 or remifentanil-4, corresponding to the target effect site concentration of this drug delivered through a TCI system. Other drugs included propofol and cisatracurium.

The paradigm exploring the baroreflex collects information continuously recorded of the RR intervals and the changes in systolic arterial pressure, before and during noxious stimuli. The hypothesis is that this paradigm explores nociception as the group with smaller doses in remifentanil will have more cardiovascular reactions in response to noxious stimuli.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I-II
* undergoing lumbar surgery for discal hernia
* body mass index <30 kg/m2

Exclusion Criteria:

* ASA classification III-IV
* cardiac history that precludes RR recording : atrial fibrillation, arterial hypertension, active cardiac pacing, chronic treatment with beta-blockers, alpha-blockers, calcium-blockers and angiotensin receptors inhibitors
* diabetes
* regular intake of cocaine, alcohol
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
changes in the baroreflex in response to noxious stimuli | intraoperative

SECONDARY OUTCOMES:
perioperative requirements in anesthetic agents. | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois PAYEN, M.D., Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France